CLINICAL TRIAL: NCT01803048
Title: A Model for Predicting Cognitive and Emotional Health From Structural and Functional Neurocircuitry Following Traumatic Brain Injury
Brief Title: Predicting Cognitive and Emotional Health From Neurocircuitry Following TBI
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, William D. Killgore, Principal Investigator, University of Arizona
Other Study IDs: 1407388572
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Diffusion Weighted Imaging; Resting State Functional Connectivity; Cognition
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- TBI: 30 individuals who will be tested at two weeks post-TBI; 30 individuals who will be tested at one month post-TBI; 30 individuals who will be tested at three months post-TBI; 30 individuals who will be tested at six months post-TBI; 30 individuals who will be tested at 12 months post-TBI.
- Healthy Control: 30 healthy individuals with no history of TBI

SUMMARY:
Abnormalities in structural and functional connectivity between brain regions have been suggested as putative biomarkers of mild traumatic brain injury (TBI) and significant contributors to neuropsychological functioning and injury outcome. The purpose of this study is to use two advanced magnetic resonance imaging (MRI) techniques called diffusion-weighted imaging (DWI) and resting state functional MRI to compare structural and functional connectivity between individuals with documented mild TBI and healthy controls. To evaluate the significance of structural and functional connectivity for behavior, the brain imaging data will then be related to measures of cognition and emotion. Over a 4-year period, 150 adults with documented mild TBI and 30 healthy controls will participate in the study.

The study will investigate the following questions and hypotheses:

1. Evaluate the DWI metric fractional anisotropy (FA) as a measure of white matter integrity across multiple stages of recovery following mild TBI relative to healthy controls. It is hypothesized that mild TBI will be associated with greater white matter abnormalities than healthy controls.
2. It is hypothesized that there will be a relationship between FA, cognition and emotion as a function of the injury.
3. It is hypothesized that functional connectivity will be related to FA.

ELIGIBILITY:
Inclusion Criteria:

* English as first language
* Ability to provide informed consent
* For TBI group: documented TBI experienced within 12 months prior to testing.

Exclusion Criteria:

* Metal within the body, claustrophobia or other contraindications for MRI
* Complicating medical conditions that may influence the outcome of neuropsychological assessment or neuroimaging (e.g., HIV, brain tumor, etc.)
* Less than 9th grade education
* History of alcoholism or substance use disorder
* Excess current alcohol use or illicit substance use
* for Healthy Controls (HC): life-time history of TBI or Axis I disorder
* Pregnancy (ruled out by urine β-HCG)
* Colorblindness
* for HC: Having participated in a sport with a high risk of concussive/subconcussive blows for a period of at least 1 month including but not limited to: football, rugby, boxing, ice hockey, wrestling, soccer, martial arts

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: One hundred eighty participants aged 20-45, including 150 adults with documented mild TBI and 30 healthy controls (HC) will participate in this study. Participants in the TBI group will include 30 individuals who will be tested at two weeks post-TBI; 30 individuals who will be tested at one month post-TBI; 30 individuals who will be tested at three months post-TBI; 30 individuals who will be tested at six months post-TBI; and 30 individuals who will be tested at 12 months post-TBI. Participants will be recruited from the local area of Boston, MA, via IRB-approved flyers and advertisements placed in newspapers, on the radio and within vehicles of the local public transport system (e.g. buses and subway cars).
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Diffusion Weighted Imaging Metric: fractional anisotropy (FA) | Measured on the day of the MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: William D Killgore, Ph.D., Principal Investigator — University of Arizona Psychiatry Department
Locations (1):
- University of Arizona Psychiatry Department, Tucson, Arizona, United States